CLINICAL TRIAL: NCT03994497
Title: Evaluation of the Level of Expression of CD45RC on T Lymphocytes as a Predictive Biomarker of Acute Rejection After Renal Transplantation
Acronym: ECLAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 49RC18_0018
Record Dates: First submitted 2019-06-11; First posted 2019-06-21 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient in need of a kidney transplant (Other)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples the day of the surgery and 4 times during the next year. Blood samples and histological slides taken at each biopsy and if there is suspicion of rejection of the graft

SUMMARY:
Chronic renal failure is a major public health problem in industrialized countries, due to its frequency - about 3 million patients in France - and its socio-economic impact. At the end stage of renal failure, renal transplantation is the best treatment, allowing an improvement in patient survival compared to treatment by extra-renal purification. Despite improved immunosuppressive strategies, allograft rejection is common in transplantation - between 15% and 25% in the first year - and is associated with lower renal graft survival.

Different risk factors for rejection have been well identified, such as the young age of the recipient or a high number of human leukocyte antigen (HLA) incompatibilities between the donor and the recipient. However, these risk factors do not accurately identify the risk of acute rejection in order to optimize and individualize immunosuppressive strategies.

Also, the search for biomarkers to predict allograft tolerance prior to transplant is a major goal in renal transplantation.

The onset of acute rejection is caused by the ability of the recipient's T cells to recognize alloantigens. The CD45 molecule is a highly expressed tyrosine phosphatase on the surface of the lymphocytes that plays an important role in the activation of the T cell.

Investigators showed that the level of expression of CD45RC on T lymphocytes was associated with the risk of acute rejection. Thus, from a retrospective cohort of 89 renal transplant patients followed, recipients with a high percentage of circulating CD8 lymphocytes expressing high CD45RC (CD45RChigh) before transplant had a 5 to 8-fold higher risk of developing acute rejection of allograft during follow-up (11-year average follow-up) compared to recipients with a low percentage of CD8+CD45RChigh.

The purpose of this study is to confirm the first retrospective results on a larger prospective and contemporary regional cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 70 years old
* Patients in care for a first priority renal transplant.
* Patients with low immunological risk
* Patients with prior written informed consent

Exclusion Criteria:

* Poor understanding of the French language
* Pregnant, breastfeeding or partying women
* Persons deprived of liberty by an administrative or judicial decision
* Persons undergoing psychiatric care under duress
* Adults who are subject to a legal or non-state protection measure to express their consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of patient with acute rejection diagnosis confirmed by anatomopathological analysis of a graft biopsy | 12 months

SECONDARY OUTCOMES:
Rate of CD45RC for patient with acute rejection suspicion | 12 months
  acute rejection confirmed or not
Rate of CD45RC on circulating T lymphocytes | from date of randomization until the date of acute rejection, up to 12 months
  Evolution of the expression of CD45RC in the first year after introduction of immunosuppressive therapy
Rate of CD45RC on circulating T lymphocytes the day of acute rejection | 12 months
  day of acute rejection
Rate of CD4, CD8, CD45RA, CD25, CD127, CD19 markers on T cells the day of acute rejection | 12 months
  day of acute rejection
anti-HLA antibodies' dosage at the time of acute rejection | 12 months
cytokines' dosage | Day 1
  describe cytokine profile

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Anne-Sophie GARNIER, Angers, France